CLINICAL TRIAL: NCT03212885
Title: Deep Brain Stimulation (DBS) of the Rostral Zona Incerta (rZI) for Parkinson's Disease (PD): Clinical Efficacy and Evaluation of Adverse Effects
Brief Title: Stimulation of the Rostral Zona Incerta for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1443
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 (Experimental): STN Monopolar Stimulation
  Interventions: Device: Deep Brain Stimulation
- 2 (Experimental): rZI + STN stimulation
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Electrode that provides electrical stimulation to deep brain structures for relief of Parkinson's Disease symptoms.

SUMMARY:
Patients with Parkinson's Disease who undergo Deep Brain Stimulation surgery receive symptom relief due to electrical stimulation of the brain. The target for the stimulation, in many cases, is the subthalamic nucleus (STN). The brain area just above the STN is called the rostral Zona Incerta (rZI). The rZI may be a potential target for deep brain stimulation, in combination with the STN.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of an area of the brain called the subthalamic nucleus (STN) is an effective treatment in Parkinson's disease (PD). However, stimulating the STN can lead to unwanted side effects that involve muscle movements (dyskinesias) and behavior and mood problems. DBS of a different brain structure, called the rostral zona incerta (rZI), has been demonstrated to be as effective as stimulating the STN, without any unwanted side effects in several studies. However, there is great variability in reported efficacy and adverse effects of rZI stimulation likely due to challenges in locating this area in the brain. The goals of this study are 1) to develop an improved method for targeting the rZI 2) determine efficacy of rZI with STN stimulation compared with STN stimulation alone, 3) evaluate any stimulation adverse effects of combined stimulation of the rZI and STN.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease,
* No current deep brain stimulating electrodes

Exclusion Criteria:

* Other movement disorders,
* Parkinson's Disease with already implanted electrode.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Motor testing | 1 week
  Blinded UPDRS testing

SECONDARY OUTCOMES:
Dyskinesias | 1 week
  Unified Dyskinesia Rating Scale
Cognition | 1 week
  Montreal Cognitive Assessment
Depression | 1 week
  Hamilton Depression Rating Scale
Anxiety | 1 week
  Hamilton Anxiety Rating Scale
Suicide | 1 week
  Columbia Suicide Severity Ratting Scale
Non-motor features of Parkinson's disease | 1 week
  Movement Disorder Society-UPDRS I
Motor aspects of daily living | 1 week
  Movement Disorder Society-UPDRS II

CONTACTS AND LOCATIONS:
Overall Officials: Drew S Kern, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No